CLINICAL TRIAL: NCT01148953
Title: A Phase 1, Randomized, Single-Blind, Placebo-Controlled, Dose Escalation Trial to Evaluate the Safety and Tolerability of a Single Dose of Intravenous ALN-TTR01 in Patients With TTR Amyloidosis
Brief Title: Trial to Evaluate Safety and Tolerability of ALN-TTR01 in Transthyretin (TTR) Amyloidosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALN-TTR01-001; 2009-017383-16 (EudraCT Number)
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Transthyretin Mediated Amyloidosis (ATTR)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALN-TTR01 (Active Comparator)
  Interventions: Drug: ALN-TTR01
- Sterile Normal Saline (0.9% NaCl) (Placebo Comparator)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: ALN-TTR01 — Dose levels between 0.01 and 1.0 mg/kg by intravenous (IV) infusion
  Arms: ALN-TTR01
Drug: Sterile Normal Saline (0.9% NaCl) — Calculated volume to match active comparator
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of a single dose of ALN-TTR01 in patients with transthyretin (TTR) mediated amyloidosis (ATTR).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of TTR amyloidosis
* Adequate blood counts, liver and renal function
* Women of child-bearing potential must have a negative pregnancy test, cannot be breast feeding, and must use an adequate method of birth control
* Males agree to use appropriate contraception
* Willing and able to comply with protocol-required visit schedule and visit requirements and provide written informed consent.

Exclusion Criteria:

* Known human immunodeficiency virus (HIV) positive status
* Receiving antibiotics for bacterial infection within 7 days of screening
* Known or suspected systemic viral, parasitic or fungal infection
* Receiving an investigational agent within 30 days prior to study drug administration
* Poor cardiac function
* Considered unfit for the study by the Principal Investigator
* Known sensitivity to oligonucleotides
* Employee or family member of the sponsor or the clinical study site personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The proportion of patients experiencing adverse events (AEs), serious adverse events (SAEs), and study drug discontinuation. | Up to 28 Days

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ALN-TTR01 (Cmax, tmax, t1/2, AUC0-last, CL) | Up to 70 days
Effect of ALN-TTR01 on Circulating TTR Levels (Determination of % Lowering of TTR to Pretreatment/Baseline TTR Level) | up to 70 days

CONTACTS AND LOCATIONS:
Overall Officials: Jared Gollob, MD, Study Director — Alnylam Pharmaceuticals Inc
Locations (4):
- Clinical Site, Le Kremlin-Bicêtre, France
- Clinical Site, Porto, Portugal
- Clinical Site, Umeå, Sweden
- Clinical Site, London, United Kingdom

REFERENCES:
- [Derived] Coelho T, Adams D, Silva A, Lozeron P, Hawkins PN, Mant T, Perez J, Chiesa J, Warrington S, Tranter E, Munisamy M, Falzone R, Harrop J, Cehelsky J, Bettencourt BR, Geissler M, Butler JS, Sehgal A, Meyers RE, Chen Q, Borland T, Hutabarat RM, Clausen VA, Alvarez R, Fitzgerald K, Gamba-Vitalo C, Nochur SV, Vaishnaw AK, Sah DW, Gollob JA, Suhr OB. Safety and efficacy of RNAi therapy for transthyretin amyloidosis. N Engl J Med. 2013 Aug 29;369(9):819-29. doi: 10.1056/NEJMoa1208760. PMID 23984729